CLINICAL TRIAL: NCT03946501
Title: Clinical Research and Data Collection During the Investigation: Influence of a Dedicated Staff
Acronym: CRA-MD
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2018Ao003
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Clinical Research Inclusion
Keywords: missing data; clinical research; clinical research assistant
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- clinical research visit
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
The aim of the study was to evaluate the interest of the recourse of a staff dedicated as CRA to data collection in clinical research

DETAILED DESCRIPTION:
Objectives of clinical studies are notably to evaluate new therapies, to improve diagnostic techniques, to make medico-economic decisions and to enrich scientific knowledge. Clinical studies findings can influence medical practice, or even motivate decisions by public health authorities. The rigor in their behavior is therefore an imperative to respect.

Thus, the quality of the data collected is essential. However, even if the reliability of the clinical data is guaranteed by the monitoring, the completeness of the data remains exceptional.

The increase of data required in clinical studies has led to the emergence of a specialized staff to assist investigators: the clinical research assistants. With dedicated time and specialization in data collection, they facilitate the conduct of clinical studies. However, this data collection aid has not been evaluated.

ELIGIBILITY:
Inclusion Criteria:

- clinical research visit performed in Reims university hospital between January 2010 and January 2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical research visit performed in Reims university hospital, with or without the help of a clinical research assistant
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Missing data | Day 0
  Data was considered missing because of its absence when finalizing the data

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Ghenim S, Feron T, Barbe C, Wolak-Thierry A, Jolly D. [Clinical research and data collection during the investigation: Influence of a dedicated staff]. Therapie. 2018 May-Jun;73(3):267-272. doi: 10.1016/j.therap.2017.10.003. Epub 2017 Nov 11. French. PMID 29198734